CLINICAL TRIAL: NCT06124911
Title: Comparison of Two Low-dose Resistance Training Modalities on Strength, Functional Capacity, and Quality-of-life in Healthy, Community-dwelling, Untrained Older Adults: a Randomised Controlled Trial
Brief Title: Low-dose Maximal-intent Versus Controlled-tempo Resistance Training on Quality-of-life in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU2863
Record Dates: First submitted 2023-10-29; First posted 2023-11-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2023-11

CONDITIONS: Quality of Life
Keywords: Activities of Daily Living; Balance; Independence; Mobility; Untrained

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Maximal-intent Resistance Training - 3x5 (MI3x5) (Experimental): The max-intent group were instructed and encouraged to deliberately commit to exerting maximal effort and force during the concentric phase of the leg press with the intention of achieving the greatest velocity possible. This group completed 3 sets of 5 repetitions at 60% one-repetition maximum.
  Interventions: Other: Leg Press Resistance Training (3x5)
- Maximal-intent Resistance Training - 5x5 (MI5x5) (Experimental): The max-intent group were instructed and encouraged to deliberately commit to exerting maximal effort and force during the concentric phase of the leg press with the intention of achieving the greatest velocity possible. This group completed 5 sets of 5 repetitions at 60% one-repetition maximum.
  Interventions: Other: Leg Press Resistance Training (5x5)
- Controlled-tempo Resistance Training - 3x5 (CT3x5) (Experimental): The controlled-tempo group followed a metronome for both eccentric and concentric phases of the leg press with the intention of maintaining a steady three-second concentric and three-second eccentric. This group completed 3 sets of 5 repetitions at 60% one-repetition maximum.
  Interventions: Other: Leg Press Resistance Training (3x5)
- Controlled-tempo Resistance Training - 5x5 (CT5x5) (Experimental): The controlled-tempo group followed a metronome for both eccentric and concentric phases of the leg press with the intention of maintaining a steady three-second concentric and three-second eccentric. This group completed 5 sets of 5 repetitions at 60% one-repetition maximum.
  Interventions: Other: Leg Press Resistance Training (5x5)

INTERVENTIONS:
Other: Leg Press Resistance Training (3x5) — Leg Press resistance training at 60% one-rep-max for three sets of five repetitions
  Arms: Controlled-tempo Resistance Training - 3x5 (CT3x5); Maximal-intent Resistance Training - 3x5 (MI3x5)
Other: Leg Press Resistance Training (5x5) — Leg Press resistance training at 60% one-rep-max for five sets of five repetitions
  Arms: Controlled-tempo Resistance Training - 5x5 (CT5x5); Maximal-intent Resistance Training - 5x5 (MI5x5)

SUMMARY:
The aims of this study were to:

1. Compare the effects of low-dose Maximal Intent and Controlled Tempo Resistance Training on untrained healthy older adults' quality-of-life, functional capacity, and strength.
2. Qualitatively explore perceptions of Maximal Intent and Controlled Tempo Resistance Training in older adults.

Older adults are defined as being 60 or more years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were between 30-60 years old
* Uninjured
* Had no cardiovascular or neuromuscular conditions
* Had not participated in lower-limb resistance training in the previous six months.

Exclusion Criteria:

* Participants were excluded if they had either taken part in any lower-limb resistance training in the last six months
* Had underlying health condition(s) that prevented them from participating in resistance training
* Regularly met or exceeded the UK recommended physical activity guideline of 150-minutes of moderate to intense physical activity per week.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Quality-of-life | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Participant quality of life (measured through focus group questions & SF-36)

SECONDARY OUTCOMES:
Balance | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Using the biodex to do a 3 x 20s double-foot eyes-open balance test on Level 6.
6-minute Walk Test | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  A "brisk"-paced 6-minute walk test.
Timed-up-and-go | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Standing from a chair, walking to a point 3 metres away, turn, and return to the chair as quick as possible whilst walking.
30-second sit-to-stand (30s-Sit-to-Stand) | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Maximal amount of repetitions a participant can stand up from a chair in 30-seconds.
Strength | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Participants one-repetition max on leg press machine.
Body Mass Index | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Mass and height will be combined to report BMI in kg/m^2
Strength-to-mass Ratio | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Mass and Leg Press 1RM will be combined to calculate strength-to-mass ratio.
Leg press one-rep-max velocity pre-to-post | At baseline and Week 1, mid (Week 4), and post (Week 9), out of a total study duration of 9 weeks.
  Velocity (m/s) of leg press measured at post-intervention, using baseline one-rep-max.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson LT, Behm DG, Goodall S, Mason R, Stuart S, Barry G. Effects of maximal-versus submaximal-intent resistance training on functional capacity and strength in community-dwelling older adults: a systematic review and meta-analysis. BMC Sports Sci Med Rehabil. 2022 Jul 16;14(1):129. doi: 10.1186/s13102-022-00526-x. PMID 35842655